CLINICAL TRIAL: NCT04125355
Title: Care to Caregiver: The Effect of Reflexology on Sleep and Anxiety of Cancer Caregiver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, İsmail TOYGAR, Research Assistant, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EgeHemsirelik
Record Dates: First submitted 2019-09-30; First posted 2019-10-14 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Sleep; Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo control
  Interventions: Other: Placebo
- Reflexology (Experimental): foot reflexology
  Interventions: Other: Reflexology

INTERVENTIONS:
Other: Reflexology — Foot reflexology massage for 3 consecutive days and 60 minutes per day.
  Arms: Reflexology
Other: Placebo — Placebo for 3 consecutive days and 60 minutes per day. This intervention only include touch to the foot, it doesn't include deep stimulation.
  Other Names: plasebo
  Arms: Placebo

SUMMARY:
Introduction and Aim: With the increase in life expectancy in cancer, it gains importance in the care process and the problems experienced by caregivers. However, the problems experienced by individuals caring for cancer patients are often ignored. The most common problems faced by cancer caregivers are sadness, anxiety, sleep disorders, and fatigue. Although reflexology has positive effects on sleep and anxiety in different patient groups, there is no study on its effectiveness in cancer caregivers. The aim of this study was to evaluate the effectiveness of reflexology on sleep and anxiety of caregivers.

Materials and Methods: The study was conducted as a double-blind placebo-controlled design. After the groups were determined with block randomization, the reflexology investigation was applied to the experimental group for three consecutive days, while for the placebo group, the hands was moved around the foot for the same periods but no deep stimulation was applied. On the fourth day, a sociodemographic diagnostic form, state anxiety scale and Richard-Campbell Sleep Scale were administered to the participants by a blinded researcher. Data were analyzed with SPSS 25.0 package program. Written permission was obtained from the relevant ethics committee, hospital and participants to conduct the study.

DETAILED DESCRIPTION:
Introduction and Aim: With the increase in life expectancy in cancer, it gains importance in the care process and the problems experienced by caregivers. However, the problems experienced by individuals caring for cancer patients are often ignored. The most common problems faced by cancer caregivers are sadness, anxiety, sleep disorders, and fatigue. Although reflexology has positive effects on sleep and anxiety in different patient groups, there is no study on its effectiveness in cancer caregivers. The aim of this study was to evaluate the effectiveness of reflexology on sleep and anxiety of caregivers.

Materials and Methods: The study was conducted as a double-blind placebo-controlled design. After the groups were determined with block randomization, the reflexology investigation was applied to the experimental group for three consecutive days, while for the placebo group, the hands were moved around the foot for the same periods but no deep stimulation was applied. On the fourth day, a sociodemographic diagnostic form, state anxiety scale, and Richard-Campbell Sleep Scale were administered to the participants by a blinded researcher. Data were analyzed with SPSS 25.0 package program. Written permission was obtained from the relevant ethics committee, hospital and participants to conduct the study.

ELIGIBILITY:
Inclusion Criteria:

* care to cancer patients at least for 6 months

Exclusion Criteria:

* decline to participate in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Sleep | 3 day
  Quality of sleep - richard campbell sleep questionnaire used to determine the quality of sleep of the patients. This questinairre used for both groups. The minimum total score in the scale is 0 and maximum is 600. The increase of the total score shows the increase the quality of sleep. the scale don't have any subscale
Anxiety | 3 day
  Level of Anxiety - The state anxiety inventory used to determine anxiety level of patients. This inventory used for both groups. The lowest total score of the scale is 20 and to highest is 80. the increase of the total points indicates the increase in anxiety. the scale don't have any subscale.

CONTACTS AND LOCATIONS:
Overall Officials: İsmail TOYGAR, Ph.D., Study Director — Ege University
Locations (1):
- Ege University Faculty of Medicine Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
undecided for now